CLINICAL TRIAL: NCT05774080
Title: An Observational Study of Patients With Chronic Gastrointestinal Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-GASTRO
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease Cohort: Observational
  Interventions: Other: Observational
- Engaged Cohort: Observational
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
TARGET-GASTRO is an observational research study to conduct a comprehensive review of outcomes for patients with the chronic gastrointestinal (GI) diseases: eosinophilic gastrointestinal disease (EGID), ulcerative colitis (UC) or Crohn's disease (CD).

ELIGIBILITY:
Disease Cohort

Inclusion Criteria:

* Adult* patients at the time of enrollment with a diagnosis or major symptom of EGIDs, UC, or CD by ICD-10 code in the EHR interface

Exclusion Criteria:

* Death
* Manual removal (sponsor or site request)
* No EHR interface encounter > 3 years.

Engaged Cohort

Inclusion Criteria:

* Adult* patients diagnosed and managed for these conditions invited to participate
* Ability to provide written informed consent

Exclusion Criteria:

* Patient expressed desire to withdraw consent to complete PROs
* Failure to complete PROs within 24 weeks of initial invitation
* Greater than 24 months lapse of survey completion after baseline surveys completed
* Additionally, the criteria detailed for Disease Cohort apply to the Engaged Cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adults who are being managed for the chronic GI diseases EGIDs, UC or CD.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2037-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
To characterize the natural history of disease in patients with GI disease from various etiologies | 20 Years
To assess safety and effectiveness of treatments | 20 Years

SECONDARY OUTCOMES:
To evaluate provider management practices in the treatment of patients with EGIDs, UC and CD | 20 Years
To evaluate longitudinal and patient reported outcomes in patients with EGIDs, UC and CD | 20 Years
To select and evaluate quality of care measures for patients with GI Diseases | 20 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Atrium Health/Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided